CLINICAL TRIAL: NCT02717520
Title: Long Term Clinical Evaluation of a Posterior Glass Hybrid System vs. Composite Resin: a Controlled Clinical MultiCenter Study
Brief Title: Long Term Clinical Evaluation of a Posterior Glass Hybrid System vs. Composite Resin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zagreb (Other)
Collaborators: University of Milan (Other); University of Belgrade (Other); Ege University (Other)
Responsible Party: Principal Investigator, Ivana Miletic, Professor, University of Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-PA-26-7/2015
Record Dates: First submitted 2016-03-08; First posted 2016-03-23 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Dental Restoration
Keywords: glass hybrid; composite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All study participants (Experimental): One permanent molar with an approximal and occlusal carious lesion restored with EQUIA Forte, and one permanent molar with an approximal and occlusal carious lesion restored with Tetric EvoCeram
  Interventions: Device: EQUIA Forte and Tetric EvoCeram

INTERVENTIONS:
Device: EQUIA Forte and Tetric EvoCeram — GC cavity conditioner (20% polyacrylic acid) will be applied for 10 sec, rinsed and the cavity will be dried with a cotton pellet. EQUIA Forte will be prepared according to the manufacturer instructions, applied in bulk and compacted with a condenser. The self-curing restoration will be finished after hardening, approximately 2 min 30 sec after the start of the capsule mixing, using Arkansas stones under water cooling. EQUIA Forte Coat will be applied to the surfaces and light cured with D-light for 20 sec.
  Enamel will be etched with 37% orthophosphoric acid for 10 sec. After the acid gel removal, the cavity will be carefully dried. The adhesive (Adhese 2, Ivoclar Vivadent) will be applied and light cured with D-light (1200 mW/cm2, slow mode) for 10 sec. The composite resin will be placed with an incremental technique (2 mm layers), and light-cured with D-light (20 sec). Restorations will be finished with fine diamond and carbide burs in slow and high-speed hand-piece and polished.

SUMMARY:
The primary objective of this study is to evaluate long-term clinical performance of a glass hybrid restorative system (glass-ionomer) vs. composite resin material over a period of five years. The secondary objective is to evaluate the suitability of intraoral impressions for the assessment of wear of teeth and restorative materials over five years. For that purpose the replica method and scanning 3-D laser equipment and matching software will be used.

The first null hypothesis is that there would be no difference in clinical performance between restorative materials after five years. The second null hypothesis is that wear between the restorative materials will be the same after five years.

This is a multicentre, controlled clinical study conducted in Croatia, Italy, Turkey and Serbia. Eligible participants are all adults aged 18 or over with indication of restorative treatment on vital teeth in posterior molar region, limited to two surface in a healthy subjects. Exclusion criteria are presence of full dentures or crowns and bridges in occlusal contact with teeth indicated for restorative treatment, severe bruxing and unstable physiological or medical health, pregnancy and lactation, radiation therapy or using drugs. Each patient is receiving two restorative treatment (GIC-EQUIA Forte and composite resin material Tetric EvoCeram) each of which will be localized on molar teeth on either side of the mouth. Two independent examiners will evaluate the restorations at each site one week after placement and at one, two, three, four and five years according to the FDI criteria. After, three and five years recall, impressions of both restorations is taken and the casts is analysed by a 3D laser scanner.

DETAILED DESCRIPTION:
Tooth vitality will be confirmed with cold test (ethyl chloride) and registrated. Bleeding of the gingiva will be recorded using a periodontal probe. Local anesthesia will be applied to prevent pain and discomfort during cavity preparation. Tooth surface will be cleaned using a commercial non fluoride prophy paste (Cleanic, fluoride free, Kerr dental). The cavity preparations will be performed by removing old fillings or/and opening carious lesions using rounded and cylindric diamond burs (Komet). Round tungsten carbide burs (Komet) and hand instruments will be used to excavate carious dentine in both groups. For composite resin restoration, sound dentin verification will be based on probing and tactile sensation. No marginal bevel will be prepared and a horizontal platform (avoid apical shift) in approximal box will be made. Before placement of the materials, impressions will be taken to registrate cavity depth.

Restorations with EQUIA Forte (GC corp., Tokyo, Japan) will be placed according to the manufacturer recommendations. The site will be isolated with cotton rolls. A sectional metal matrix system and wedge will be placed. GC cavity conditioner (20% polyacrylic acid, GC) will be applied for 10 sec., rinsed and the cavity will be dried with a cotton pellet. EQUIA Forte (GC) will be prepared according to the manufacturer instructions, applied in bulk and compacted with a condenser. The self-curing restoration will be finished after hardening, approximately 2 minutes 30 seconds after the start of the capsule mixing, using Arkansas stones under water cooling. Occlusion and articulation will be checked by using two sided and coloured articulating paper (blue for occlusion and red for articulation) 20 microns thickness. EQUIA Forte restoration will be rinsed and gently dried. EQUIA Forte Coat (GC) will be applied to the surfaces using a micro-tip applicator. The coated surface will be light cured with D-light (GC) for 20 seconds. Patients will be instructed not to eat during one hour after the restoration placement.

For composite resin restoration, rubber-dam will be applied, and the same matrix system will be used. Enamel will be etched with 37% orthophosphoric acid (Ivoclar Vivadent, Schaan, Liechtenstein) for 10 sec., avoiding etching dentine as much as possible. The acid gel will be rinsed with air-water spray and the cavity will be carefully dried with a mild stream of air until the etched enamel appears white-frosted and dentin dull (avoiding to over-dry of dentine surface). The adhesive (Adhese 2, Ivoclar Vivadent) will be applied according to the manufacturer's instruction and light cured with D-light (GC, 1200 mW/cm2, slow mode) for 10 sec. The composite resin (Tetric EvoCeram, Ivoclar Vivadent) will be placed with an incremental technique (2 mm layers). Composite will be light-cured with D-light (20 sec) from the occlusal direction by placing the light tip as close as possible to the restoration. After removing of matrix, additional light curing will be performed from vestibular and palatal/lingual direction. Finishing will be performed using diamond burs. Restorations will be finished with fine diamond burs in high-speed hand-piece for gross finishing (Komet) followed by fine carbide burs in slow speed hand-piece for fine finishing (Komet). Occlusion and articulation will be checked by using two sided and coloured articulating paper (blue and red) 20 microns of thickness. Polishing will be performed using flexible polishing discs (Komet), rubber points (Compo system, Komet) with a diamond particle paste (1μm) (Gradia diapolisher). Fine polishing stripes will be used for proximal surface below the contact point.

One week after the placement of the restorations, baseline evaluation will be performed and follow-up evaluations will be done on yearly bases up to five years. Two experienced, blinded, calibrated examiners (e-calib) who will not perform clinical procedures will evaluate the restorations. Evaluation will be done by using loops (magnification x 2.5).

Impressions obtained before procedure, after cavity preparation, at baseline, three and five years will be directly scanned using 3D laser scanning device (GC Aadva Lab scan). After direct impression scanning, a gypsum cast (GC Fujirock EP OptiXscan) will be also made (baseline, three and five years). These models will be scanned for wear analysis with the GC Aadva software in order to compare two different evaluation methods.

At baseline and at every recall, four photos will be taken: one photo from the occlusal view, buccal view, oral view and direct view.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with indication for restorative treatment on vital teeth in posterior molar region
* Restorations limited to two surfaces with one proximal cavity in occlusion
* Favourable and stable occlusal relationship between the remaining teeth.

Exclusion Criteria:

* Subject with full dentures or crowns and bridges in occlusal contact with teeth indicated for restorative treatment
* Subject has a history of drug abuse, addiction to medication or alcohol abuse within the previous year
* Pulp exposure
* Allergy to any ingredient of a material
* Severe bruxing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-09; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evaluating surface and marginal staining of the materials | 5 year
  Criteria established by Hickel et al. (2007) will be used
Evaluating fracture and retention of the materials | 5 year
  Criteria established by Hickel et al. (2007) will be used
Evaluating marginal adaptation and discoloration of the materials | 5 years
  Criteria established by Hickel et al. (2007) will be used
Evaluating wear of the materials | 5 years
  Criteria established by Hickel et al. (2007) will be used

SECONDARY OUTCOMES:
Evaluating suitability of direct impression scanning vs. replica model scanning for wear assessment | 5 years
  Impressions obtained before procedure, after cavity preparation, at baseline, three and five years will be directly scanned using 3D laser scanning device (GC Aadva Lab scan). After direct impression scanning, a gypsum cast (GC Fujirock EP OptiXscan) will be also made (baseline, three and five years). These models will be scanned for wear analysis with the GC Aadva software in order to compare two different evaluation methods.

CONTACTS AND LOCATIONS:
Locations (4):
- School of Dental Medicine, Zagreb, Croatia
- Dental School, Milan, Italy
- Faculty of Dental Medicine, Belgrade, Serbia
- Ege University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Science Committee Project 2/98--FDI World Dental Federation study design (Part I) and criteria for evaluation (Part II) of direct and indirect restorations including onlays and partial crowns. J Adhes Dent. 2007;9 Suppl 1:121-47. PMID 18341239
- [Derived] Schwendicke F, Rossi JG, Krois J, Basso M, Peric T, Turkun LS, Miletic I. Cost-effectiveness of glass hybrid versus composite in a multi-country randomized trial. J Dent. 2021 Apr;107:103614. doi: 10.1016/j.jdent.2021.103614. Epub 2021 Feb 19. PMID 33617942

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT02717520/Prot_SAP_000.pdf